CLINICAL TRIAL: NCT03657979
Title: Transversus Abdominis Plane (TAP) Block in Open Abdominal Aortic Surgery : Randomized Controlled Doubled-blind Trial Comparing Ropivacaine 0.2% Versus Placebo
Brief Title: TAP-Block in Abdominal Aortic Surgery
Acronym: TAP-CACAO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Eric STEINMETZ, Professor, Centre Hospitalier Universitaire Dijon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-002355-34
Record Dates: First submitted 2018-06-29; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: analgesia; TAP-block
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental): Conventional PCA morphine +TAP-block ropivacaine 0.2%
  Interventions: Drug: Ropivacaine
- TAP-block with placebo (Placebo Comparator): Conventional PCA morphine treatment with TAP-block with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine — TAP-block Ropivacaine 0.2% during 48 hours
  Arms: Ropivacaine
Drug: Placebo — TAP-block with placebo
  Arms: TAP-block with placebo

SUMMARY:
The primary outcome of this study was the evaluation of the efficacy of TAP block on pain intensity following open abdominal aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Open abdominal aortic surgery (aneurysm or aortobifemoral bypass)
* Person who has given his written consent

Exclusion Criteria:

* Emergency surgery
* Patient with infection
* Use of opioids in the long term
* History of chronic pain
* Higher functions incompatible with the functioning of the PCA
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2012-08-29 (Actual); Study Completion 2012-08-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of morphine consumption at 24 postoperative hours | 24 hours
  Morphine consumption (Patient Controlled Analgesia) statement during the first 24 postoperative hours

SECONDARY OUTCOMES:
Evaluation of Visual Analogue Scale scores at 24 postoperative hours | 24 hours
  Visual Analogue Scale scores statement during the first 24 postoperative hours (minimum pain 0 - maximum pain 10)

CONTACTS AND LOCATIONS:
Overall Officials: Claude GIRARD, Professor, Principal Investigator — Anesthesia unit; Eric STEINMETZ, Professor, Principal Investigator — Cardiovascular and thoracic surgery unit
Locations (1):
- Cardiovascular and thoracic surgery unit, CHU Dijon, Dijon, France